CLINICAL TRIAL: NCT03914196
Title: Can Ultrasound Liver Stiffness Pre-Fontan, Post-Fontan, or Change Over Time Predict Onset and Severity of Fontan-Related Complications, Including Fontan-Associated Liver Disease
Brief Title: Fontan Associated Liver Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-7816
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Fontans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Liver Stiffness Ultrasound — Research imaging will include liver assessments of stiffness (ultrasound shear wave elastography), tissue attenuation (if available), and blood flow (gray-scale and Doppler imaging).
  Other Names: shear wave elastography (also called ARFI)

SUMMARY:
Fontan-associated liver disease (FALD), including the development of cardiac cirrhosis and liver neoplasms (benign and malignant), occurs in a majority of patients with congenital heart disease palliated with the Fontan operation. However, the specific phenotype (fibrosis only, fibrosis + lesions, etc.) of disease and severity/timing of onset are variable. Chronic passive congestion of the liver due to the absence of a functional sub-pulmonary ventricle and resultant chronic central venous hypertension is suspected to be one of the chief drivers of FALD and recent work has demonstrated that ultrasound shear wave elastography can be used to noninvasively detect and measure the degree of liver congestion. Chronic passive congestion of the liver may also be a predictor of other Fontan-related complications, such as protein losing enteropathy, plastic bronchitis, and intractable ascites.

ELIGIBILITY:
Inclusion Criteria:

1. Single ventricle physiology congenital heart disease undergoing Fontan operation;
2. ≤5 years of age at the time of stage 3 Fontan operation;
3. Ability to return for follow-up imaging.

Exclusion Criteria:

1. Inability to undergo ultrasound imaging.
2. Non-English speaking patients, as breath-hold is required for US shear wave elastography in older children due to excursion of the liver with breathing.

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients that are undergoing a Fontan Palliation during cardiothoracic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre/Post Fontan Liver Stiffness Changes | 5 years
  to determine if there are differences between patients with regard to liver stiffness (hepatic congestion) pre- and post-Fontan operation or with regard to change in liver stiffness over time. This information will be used to drive future hypothesis-driven research related to predicting Fontan-related outcomes based on measured liver stiffness.

SECONDARY OUTCOMES:
Correlate liver stiffness measurements with clinical outcomes at 3-, 5-, and 10-years post stage 3 Fontan operation | 10 years
  1. Time to anatomic Fontan pathway obstruction or physiologically high resistance, need for Fontan pathway intervention, need for cardiac transplant evaluation or actual transplantation, and need for mechanical cardiac support evaluation or actual implementation (e.g., ventricular assist device)
  2. Lymphatic abnormalities (e.g., protein losing enteropathy, plastic bronchitis, intractable ascites)
  3. FALD
  i. MRI outcomes (e.g., increased liver stiffness [do US and MRI measures of liver stiffness correlate?], portal hypertension, development of focal liver lesions) ii. Liver laboratory assessments (e.g., ALT, AST, bilirubin, alkaline phosphatase, GGT) iii. PELD score iv. VAST score v. Need for liver transplant evaluation or actual transplantation d. Available biopsy (liver and cardiac) data e. Available cardiac catheterization data f. Available cardiac echocardiography and/or cardiac MRI data

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] DiPaola FW, Schumacher KR, Goldberg CS, Friedland-Little J, Parameswaran A, Dillman JR. Effect of Fontan operation on liver stiffness in children with single ventricle physiology. Eur Radiol. 2017 Jun;27(6):2434-2442. doi: 10.1007/s00330-016-4614-x. Epub 2016 Oct 17. PMID 27752831